CLINICAL TRIAL: NCT00147524
Title: Multicenter, Open-Label (Non-Comparative) Study To Evaluate Changes In Flow Mediated Dilatation During And After A 6 Months Treatment Period With Step By Step Increased Doses With Quinapril Therapy In Post-Menopausal Women With Mild Or Moderate Hypertension
Brief Title: Non-Comparative Study To Evaluate Changes In FMD After Quinapril Therapy In Hypertensive Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A9061010
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2007-04-30 (Estimated); Status verified 2007-04

CONDITIONS: Menopause; Hypertension
MeSH Terms: conditions — Hypertension | interventions — Quinapril

INTERVENTIONS:
Drug: quinapril
Procedure: Laser Doppler imaging

SUMMARY:
ACE inhibitors are thought to modify the endothelium in a number of ways. Quinapril is an effective and well-tolerated ACE-I for the treatment of patients with hypertension and congestive heart failure. Quinapril produces favourable haemodynamic changes and improves ventricular and endothelial function in patients with various cardiovascular disorders. These effects are mediated through the binding of quinaprilat to both tissue and plasma-ACE.

Quinapril 10 to 40 mg once daily improved endothelial function (as measured by improved FMD or reduced vasoconstrictive/increased vasodilative response to Ach) in patients with CAD and hypertension over 2 to 6 months of therapy; improved endothelial function was also observed in patients with CHF receiving a single infusion of quinaprilat. In general, quinapril showed neutral or beneficial effects on lipid profiles, glycaemia and renal haemodynamics. (3) There are no data available considering effects of quinapril on endothelial dysfunction in post- menopausal woman with mild to moderate hypertension and with pathological endothelial function.

ELIGIBILITY:
Inclusion Criteria:

* pathological baseline FMD (< 5%) at screening
* women in post-menopause at least for 2 years (post-menopausal defined as having amenorrhea for Å' 2 years)
* mild or moderate hypertension (BP > 140/90 mmHg)

Exclusion Criteria:

* uncontrolled severe hypertension (BP > 180/110 mmHg)

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70
Dates: Start 2003-10; Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of 10, 20 and 40 mg daily sequential quinapril doses in a 3 x 8 weeks treatment period as changes to baseline pathological FMD.

SECONDARY OUTCOMES:
1.In a subgroup of about 30 patients to assess microvascular vasomotor function by laser Doppler (LD) techniques. For all patients: 2.Evaluation of changes of BP parameters. 3.Changes in PAI-1 level. 4.Collect safety data.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- Hungary (5):
  - Pfizer Investigational Site, Hódmezővásárhely, Csongrád megye
  - Pfizer Investigational Site, Budapest
  - Pfizer Investigational Site, Mátészalka
  - Pfizer Investigational Site, Szeged
  - Pfizer Investigational Site, Szombathely